CLINICAL TRIAL: NCT04581356
Title: The Effect of Voxelotor on Exercise Capacity of Youths With Sickle Cell Anemia
Brief Title: Voxelotor Sickle Cell Exercise Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Elizabeth Yang, MD, PhD (Other)
Collaborators: Pediatrix (Other); University of California, San Francisco (Other); Global Blood Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Elizabeth Yang, MD, PhD, Pediatric Hematologist, Director, Sickle Cell Program, Pediatric Specialists of Virginia
Organization: Pediatric Specialists of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-C006
Record Dates: First submitted 2020-09-11; First posted 2020-10-09 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Intervention Model Description: single-arm, open-label, pilot study in which each subject compared to him/herself
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- voxelotor (Experimental): Voxelotor 1500mg daily orally
  Interventions: Drug: Voxelotor

INTERVENTIONS:
Drug: Voxelotor — daily voxelotor 1500mg oral medication
  Other Names: GBT440, Oxbryta

SUMMARY:
This study is a pilot, open-label, single-arm study to evaluate the effect of the sickle cell medication voxelotor on exercise capacity, as measured by cardiopulmonary exercise testing (CPET) in patients 12 years of age and older with sickle cell anemia (SCA).

DETAILED DESCRIPTION:
This study will assess exercise capacity by cardiopulmonary exercise testing (CPET) before and after 8 weeks of voxelotor therapy.

Patients with genetically severe forms of sickle cell disease, including Hgb SS, Hgb S beta 0 thalassemia, Hgb SC Harlem, etc., age 12 or older, with stable Hgb and Hgb F will be recruited. Enrolled subjects will have study labs drawn, undergo baseline CPET in the exercise lab, then take voxelotor 1500mg daily for 2 months, followed by repeat study labs and a second CPET. Each subject's CPET results before and after voxelotor will be compared, and the study labs before and after voxelotor will be compared. Each subject will be compared to him/herself.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, age > 12 years
4. In good general health as evidenced by medical history and diagnosed with a genetically severe form of sickle cell anemia (Hgb SS, Hgb S beta 0 thalassemia, Hgb SCHarlem, and others)
5. Patients who are on Hydroxyurea need to be on a stable dose for at least 3 months without anticipated change in dosing until the study is completed.
6. Ability to take oral medication and willingness to adhere to daily voxelotor and 2 CPETs at scheduled intervals.
7. For females of reproductive potential who are sexually active: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 30 days after the end of study.
8. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner

Exclusion Criteria:

1. Patients on chronic transfusions or who received a transfusion within last 8 weeks
2. Patients who had hospitalization for vaso-occlusive crisis or acute chest syndrome within 30 days prior to informed consent/assent.
3. Patients who have screening alanine aminotransferase (ALT) > 4X upper limit of normal
4. Patients who suffer from physical inactivity attributable to clinically significant musculoskeletal, cardiovascular, or respiratory comorbidities
5. Patients already taking commercially available voxelotor
6. Prior hypersensitivity to voxelotor or excipients.
7. Pregnant patients

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption (VO2) | 8 weeks
  Change in peak oxygen consumption (VO2) measured in CPET after voxelotor treatment

SECONDARY OUTCOMES:
Change in Biochemical markers of red cell sickling: Hemoglobin | 8 weeks
  Measured before and after treatment with voxelotor.
Change in Biochemical markers of red cell sickling: Reticulocyte Count | 8 weeks
  Measured before and after treatment with voxelotor.
Change in Biochemical markers of red cell sickling: Bilirubin | 8 weeks
  Measured before and after treatment with voxelotor.
Change in Biochemical markers of red cell sickling: Lactate Dehydrogenase (LDH) | 8 weeks
  Measured before and after treatment with voxelotor.
Change in Biochemical markers of red cell sickling: Haptoglobin | 8 weeks
  Measured before and after treatment with voxelotor.
Change in Biochemical markers of red cell sickling: % Fetal Hemoglobin expressing cells | 8 weeks
  Measured before and after treatment with voxelotor.
Change in Biochemical markers of red cell sickling: P50 oxygen dissociation | 8 weeks
  Measured before and after treatment with voxelotor.
Change in Biochemical markers of red cell sickling: Point of Sickling (POS) | 8 weeks
  Measured before and after treatment with voxelotor.
Change in Biochemical markers of red cell sickling: Dense Cells | 8 weeks
  Measured before and after treatment with voxelotor.

OTHER OUTCOMES:
HRQOL: Patient's Global Impression of Change (PGIC) | 8 weeks
  Health-related quality of life (HRQoL) as assessed by patient reported outcome via Patient's Global Impression of Change (PGIC) at end of treatment study visit.
  The PGIC asks patients to rate their overall improvement relative to their baseline state at the beginning of the study on a 7-point scale.
  1. No change (or condition has got worse)
  2. Almost the same, hardly any change at all
  3. A little better, but not noticeable change at all
  4. Somewhat better, but the change has not made any real difference
  5. Moderately better, and a slight but noticeable change
  6. Better, and a definite improvement that has made a real and worthwhile difference
  7. A great deal better, and a considerable improvement that has made all the difference
HRQOL: Clinical Global Impression of Change (CGIC) | 8 weeks
  Health-related quality of life (HRQoL) as assessed by clinician-reported outcome via Clinical Global Impression of Change-Improvement (CGIC-I) scale at end of treatment study visit.
  The CGIC-I is a one-item questionnaire that requires the clinician to assess how much the patient's illness has improved or worsened relative to their baseline state at the beginning of the intervention on a 7-point scale:
  1. = Very much improved
  2. = Much improved
  3. = Minimally improved
  4. = No change
  5. = Minimally worse
  6. = Much worse
  7. = Very much worse

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Yang, MD, PhD., Principal Investigator — Pediatric Specialists of Virginia; Vivian Phan, MS, Study Director — Pediatric Specialists of Virginia; Kari Wheeler, BSN, RN, Study Director — Pediatric Specialists of Virginia
Locations (1):
- Pediatric Specialist of Virginia, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Phan V, Hershenson J, Caldarera L, Larkin SK, Wheeler K, Cortez AL, Dulman R, Briere N, Lewis A, Kuypers FA, Yang E. Effect of voxelotor on cardiopulmonary testing in youths with sickle cell anemia in a pilot study. Pediatr Blood Cancer. 2023 Aug;70(8):e30423. doi: 10.1002/pbc.30423. Epub 2023 May 29. PMID 37247190

DOCUMENTS (2):
  • Study Protocol (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT04581356/Prot_000.pdf
  • Informed Consent Form (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT04581356/ICF_001.pdf